CLINICAL TRIAL: NCT01617161
Title: Prostate Advanced Radiation Technologies Investigating Quality of Life (PARTIQoL): A Phase III Randomized Clinical Trial of Proton Therapy vs IMRT for Low or Intermediate Risk Prostate Cancer
Brief Title: Proton Therapy vs. IMRT for Low or Intermediate Risk Prostate Cancer
Acronym: PARTIQoL
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: University of Pennsylvania (Other); National Cancer Institute (NCI) (NIH); Northwestern Medicine Chicago Proton Center (Unknown); ProCure Proton Therapy Center (Other); Washington University School of Medicine (Other); University of Washington (Other); Rutgers Cancer Institute of New Jersey (Other); Mayo Clinic (Other); University of Maryland, Baltimore (Other); University Hospitals Cleveland Medical Center (Other); University of Florida Proton Therapy Institute (Unknown); Provision Center for Proton Therapy (Other)
Responsible Party: Principal Investigator, Jason Efstathiou, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-497
Record Dates: First submitted 2012-06-08; First posted 2012-06-12 (Estimated); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer
Keywords: Low Risk; Intermediate Risk
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Proton Therapy; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PBT (Active Comparator): Proton Beam Therapy
  Interventions: Radiation: Proton Beam Therapy
- IMRT (Active Comparator): Intensity Modulated Radiation Therapy
  Interventions: Radiation: Intensity Modulated Radiation Therapy

INTERVENTIONS:
Radiation: Proton Beam Therapy — 5 days per week up to 9 weeks
  Arms: PBT
Radiation: Intensity Modulated Radiation Therapy — 5 times per week up to 9 weeks
  Arms: IMRT

SUMMARY:
We are studying whether men being treated for prostate cancer have the same amount of side effects from either one of two different external radiation treatments: IMRT or PBT. With IMRT, a number of x-ray beams are used to shape the radiation to the prostate. PBT is another type of external radiation treatment for prostate cancer that is used in a few centers in the United States. Protons are tiny particles with positive charge that can be controlled to travel a certain distance and stop. PBT is precise like IMRT, but it uses proton beams instead of x-ray beams.

IMRT and PBT aim to deliver most of the radiation to the prostate cancer while sparing surrounding tissues. Both IMRT and PBT have been used in the treatment of prostate cancer and are thought to be equally effective at curing prostate cancer. However, both treatments have also been shown to cause the potential side effects of radiation, including bowel, urinary and erectile problems. It is possible that side effect rates with PBT will be lower, the same, or even higher than with IMRT, but this has not been studied well to date. Though both of these radiation therapies have been used in the past to treat prostate cancer, there has never been a study that compares the effects of these two therapies to see which one has less side effects.

In this research study, we are comparing IMRT to PBT to determine which therapy best minimizes the side effects of treatment.

DETAILED DESCRIPTION:
Because no one knows which of the study options is best, you will be "randomized" into one of the study groups: IMRT or PBT. Randomization means that you are put into a group by chance, like flipping a coin. Neither you nor the research doctor will choose which group you will be in. You will have an equal chance of being placed in either group. Randomization makes the study better from a scientific point of view because it helps ensure that patients receiving IMRT and proton therapy are similar. You will be receiving only one type of radiation, either IMRT or PBT throughout your participation in the study.

Before you begin radiation therapy you will have a pelvic CT scan in order to design your radiation treatment. Doctors will use information gathered from these scans to plan the best way to deliver radiation to your tumor.

Both types of radiation therapy will be given once a day for 5 days (no weekends or holidays) for up to 9 weeks. Both IMRT and PBT will require that you lie on a table for less than 15 minutes to obtain your treatment.

During each visit you will be asked questions about your general health and specific questions about any problems that you might be having and any medications you might be taking. You will also undergo a physical exam and complete some quality of life questionnaires.

After your radiation therapy you will have follow up visits at 3,6,9,12,18,24,36,48 and 60 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with histologically confirmed adenocarcinoma of the prostate based on core-biopsy within 1 year of study entry from TRUS
* Clinical stages T1c to T2c
* PSA <20, within 6 months of study entry
* Participants who are currently receiving Dutasteride (or have received it within the last 90 days) or Finasteride (or have received it within the last 30 days) must have a PSA of ≤ 10
* Gleason score ≤6, 3 + 4 = 7, or 4 + 3 = 7
* ECOG Performance Status 0-1 as documented within 3 months prior to study entry
* Must have complete history and physical examination within 45 days of study entry and digital rectal examination of prostate within 180 days of study entry

Exclusion Criteria:

* Prior surgery (not including TURP), cryosurgery, radiofrequency ablation, chemotherapy or radiation for PCa
* Prior or planned androgen deprivation or bilateral orchiectomy
* Distant metastases, or clinically or pathologically involved lymph nodes confirmed by a CT scan within 365 days of study entry
* Hip prosthesis, inflammatory bowel disease or connective tissue disorder such as active scleroderma or lupus
* Individuals with a history of other malignancies are ineligible unless 1) they have been disease-free for at least 5 years OR 2) are deemed by the investigator to be at low risk for recurrence of that malignancy with no plans for adjuvant systemic chemotherapy and/or radiation therapy and have received overall principal investigator approval.
* Individuals who have AIDS (CD4 < 200 or an AIDS-defining illness) or are HIV positive and not on HAART therapy are ineligible.
* Major medical or psychiatric illness
* Individuals with any of the following conditions are excluded from this study:

  * Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months.
  * Transmural myocardial infarction within the last 6 months.
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration.
  * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration
  * History of Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects within the last 12 months

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 454 (Actual)
Dates: Start 2012-07-25 (Actual); Primary Completion 2025-12 (Actual); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy of PBT vs. IMRT | 2 years
  Compare the reduction in mean EPIC bowel scores for men with low or low-intermediate risk PCa treated with PBT versus IMRT at 24 months following radiation (where higher scores represent better outcomes)

SECONDARY OUTCOMES:
Disease Specific Quality of Life | 2 years
  Assess the effectiveness of PBT versus IMRT for men with low or low-intermediate risk PCa in terms of disease-specific quality of life as measured by patient-reported outcomes, perceptions of care and adverse events
Cost Effectiveness of PBT vs. IMRT | 2 years
  Assess the cost-effectiveness of PBT versus IMRT under current conditions and model future cost-effectiveness for alternative treatment delivery and cost scenarios
Radiation Dose and Bowel, Urinary and Erectile Function | 2 years
  Develop predictive models to examine the associations between selected metrics of individual radiation dose distributions and patient reported bowel, urinary and erectile function
Identification and Evaluation Biomarkers of PCa Behavior | 2 years
  Identify and evaluate biomarkers of prostate cancer behavior and response to radiotherapy
Long Term Survival | 10 years
  Assess longer-term rates of disease-specific and overall survival as well as development of late effects such as second cancers

CONTACTS AND LOCATIONS:
Overall Officials: Jason A Efstathiou, MD, DPhil, Principal Investigator — Massachusetts General Hospital
Locations (13):
- United States (13):
  - University of Florida Health Proton Therapy Institute, Jacksonville, Florida
  - Northwestern Medicine Chicago Proton Center, Chicago, Illinois
  - University of Maryland Medical Center, College Park, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mass General/North Shore Cancer Center, Danvers, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Princeton ProCure Proton Therapy Center, Somerset, New Jersey
  - University Hospital of Cleveland, Cleveland, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Provision Proton Therapy Center, Knoxville, Tennessee
  - University of Washington Medical Center, Seattle, Washington

REFERENCES:
- [Derived] Liu Y, Patel SA, Jani AB, Gillespie TW, Patel PR, Godette KD, Hershatter BW, Shelton JW, McDonald MW. Overall Survival After Treatment of Localized Prostate Cancer With Proton Beam Therapy, External-Beam Photon Therapy, or Brachytherapy. Clin Genitourin Cancer. 2021 Jun;19(3):255-266.e7. doi: 10.1016/j.clgc.2020.08.009. Epub 2020 Aug 28. PMID 32972877